CLINICAL TRIAL: NCT03800004
Title: Bone Health in Patients With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Pediatric Dermatology Research Alliance (Unknown)
Responsible Party: Principal Investigator, Megha M. Tollefson, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 17-007112
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Bone Health
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study examines the bone health in children with atopic dermatitis

DETAILED DESCRIPTION:
The goal of this study is to objectively evaluate bone health and contributing factors in children with AD. This will be compared with existing normative data. Such an objective prospective study, directly looking at bone health in children has not yet been done. This will be done using bone densitometry (DXA) and high-resolution peripheral quantitative computed tomography (HR-pQCT) for the accurate and precise measurement of bone health status. HR-pQCT is a cutting-edge technology available at only at a few academic centers in the United States that is used to measure bone strength with minimal doses of radiation. In addition, blood and urine metabolic parameters related to bone health will be analyzed, and data will be correlated with eczema severity. The results from this study will allow us to design large-scale, multi-institutional studies on bone health in this population and ultimately to guide decision making in children who may be at risk specifically regarding treatment recommendations and supportive care.

The specific aims of this project are:

1. To determine bone mineral density (BMD) and cortical and trabecular bone strength in children with atopic dermatitis, using DXA and to compare this with normative data.
2. HR-pQCT data will be compared with current known data from other diseases
3. To correlate bone mineral density with eczema severity using Eczema area and severity index (EASI) and Scoring atopic dermatitis (SCORAD) scores.
4. To determine if bone mineral density in children with atopic dermatitis correlates with bone age and bone-health specific serum markers.

ELIGIBILITY:
Inclusion Criteria:

* Children 5 to 17 years of age with a diagnosis of moderate to severe atopic dermatitis as made by a dermatologist
* Duration of atopic dermatitis symptoms for a minimum of 6 months
* Ability to cooperate with DXA and HR-pQCT procedure

Exclusion Criteria:

* Those without a confirmed diagnosis of moderate to severe atopic dermatitis
* Presence of concurrent disease that may also affect bone health, including rickets or other vitamin D deficiency, thyroid disease, renal disease, Paget's disease, osteogenesis imperfecta, inflammatory bowel disease, and other chronic inflammatory diseases
* Current use of medications that may affect bone health, including bisphosphonate, Forteo, Tymlos, denosumab, thiazide, heparin, medroxyprogesterone acetate, cyclosporine, and oral tacrolimus. However, medications that are used for atopic dermatitis treatment are allowed
* Pregnant or breast feeding females
* Inability to cooperate with the blood draw

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with a diagnosis of moderate to severe atopic dermatitis as made by a dermatologist
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Correlate bone mineral density to normative data | 2 years
  To determine bone mineral density (BMD) and cortical and trabecular bone strength in children with atopic dermatitis, using dual energy x-ray absorptiometry (DXA) and High-resolution peripheral quantitative computed tomography (HR-pQCT) and to compare this with normative data.
Correlate bone age with the Eczema area and severity index and the Scoring atopic dermatitis score | 2 years
  To correlate bone mineral density with eczema severity using Eczema area and severity index (EASI) and Scoring atopic dermatitis (SCORAD) scores
Correlate bone age with serum markers | 2 years
  To determine if bone mineral density in children with atopic dermatitis correlates with bone age and bone-health specific serum markers

CONTACTS AND LOCATIONS:
Overall Officials: Megha M Tollefson, MD, Principal Investigator — Mayo Clinic; Henry Nguyen, MD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Garg N, Silverberg JI. Association between eczema and increased fracture and bone or joint injury in adults: a US population-based study. JAMA Dermatol. 2015 Jan;151(1):33-41. doi: 10.1001/jamadermatol.2014.2098. PMID 25353616
- [Background] Haeck IM, Hamdy NA, Timmer-de Mik L, Lentjes EG, Verhaar HJ, Knol MJ, de Bruin-Weller MS, Bruijnzeel-Koomen CA. Low bone mineral density in adult patients with moderate to severe atopic dermatitis. Br J Dermatol. 2009 Dec;161(6):1248-54. doi: 10.1111/j.1365-2133.2009.09327.x. Epub 2009 Jun 4. PMID 19673879
- [Background] van Velsen SG, Knol MJ, van Eijk RL, de Vroede MA, de Wit TC, Lam MG, Haeck IM, de Bruin-Weller MS, Bruijnzeel-Koomen CA, Pasmans SG. Bone mineral density in children with moderate to severe atopic dermatitis. J Am Acad Dermatol. 2010 Nov;63(5):824-31. doi: 10.1016/j.jaad.2009.12.015. Epub 2010 Sep 17. PMID 20850893
- [Background] Wu CY, Lu YY, Lu CC, Su YF, Tsai TH, Wu CH. Osteoporosis in adult patients with atopic dermatitis: A nationwide population-based study. PLoS One. 2017 Feb 16;12(2):e0171667. doi: 10.1371/journal.pone.0171667. eCollection 2017. PMID 28207767
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials